CLINICAL TRIAL: NCT02039141
Title: Community-Based Diabetes Prevention Program for Obese Latino Youth: Every Little Step Counts
Brief Title: Diabetes Prevention Program for Obese Latino Youth
Acronym: ELSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1203007572; 5P20MD002316-07 (NIH)
Record Dates: First submitted 2013-07-31; First posted 2014-01-17 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Insulin Resistance; Diabetes
Keywords: diabetes prevention program; community based interventions; childhood obesity; insulin resistance; glucose tolerance; quality of life; Latino youth; physical activity; nutrition
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus; Pediatric Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Every Little Step Counts Intervention (Experimental): Exercise classes (3/week) Lifestyle sessions (1/week)
  Interventions: Other: Every Little Step Counts Intervention
- Delayed ELSC Intervention Group (No Intervention): Control group (delayed intervention group)

INTERVENTIONS:
Other: Every Little Step Counts Intervention — Youth participants randomized to participate in the experimental group will attend weekly healthy lifestyles education session with their parent(s)/guardian(s) and will also attend exercise sessions 3 times a week for 12 weeks. The education sessions will cover topics such as healthy eating choices, roles and responsibilities of both parents and youth in the realm of the family unit as well as in youth's own health, and self esteem among other topics. The exercise sessions will incorporate both aerobic and resistance training as well as other "free-play" physical activities i.e. basketball, volleyball etc.
  Other Names: ELSC Intervention; DPP-ELSC; ASU ELSC
  Arms: Every Little Step Counts Intervention

SUMMARY:
The purpose of this study is to examine the effects of 12 week lifestyle intervention on diabetes risk in obese Latino adolescents.

DETAILED DESCRIPTION:
Obesity in the United States has reached epidemic proportions and Latinos youth are disproportionally impacted. Pediatric obesity is associated with several chronic health conditions including insulin resistance and type 2 diabetes. However, very few interventions specifically targeting diabetes prevention for obese Latino adolescents have been developed.

Therefore, the purpose of this study is to examine the effects a culturally-grounded, community-based lifestyle intervention on psychosocial and health outcomes among obese Latino adolescents. Eligible participants of this study will be randomly selected to the intervention group or the delayed-intervention group (control group) after an initial health screening for eligibility.

Participants selected to the intervention group will attend weekly healthy lifestyle education sessions with their parent(s)/guardian(s) and three physical activity sessions / week with other youth. After which, participants will attend monthly booster group meetings for three months.

All participants will be assessed at baseline, 3 months, 6 months, and 12 months for insulin sensitivity, glucose tolerance, quality of life, fitness, and nutrition and physical activity behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Latino: self-report by parents
* Age: 14-16
* Obese: BMI percentile >= 95th percentile for age and gender or BMI >= 30 kg/m^2

Exclusion Criteria:

* Taking medication(s) or diagnosed with a condition that could influence carbohydrate metabolism, physical activity, and/or cognition
* Type 2 diabetes: Fasting plasma glucose >= 126 mg/dL or 2-hour plasma glucose >= 200 mg/dL (youth found to be diabetic through study's procedures will be referred for follow up care and excluded)
* Recent hospitalizations (previous 2 months)
* Currently enrolled in (or with in previous 6 months) a formal weight loss program
* Diagnosed depression or other condition that may impact QoL

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-08-04 (Actual)

PRIMARY OUTCOMES:
Change in Insulin Sensitivity / Glucose Tolerance, Measured at Baseline, Change 3-months, 6-months, and 12-months | Baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  Proximal indicator of diabetes risk
Change in Quality of Life Measured at Baseline, 3-months, 6-months, and 12-months | Baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  Generic and weight-specific quality of life

SECONDARY OUTCOMES:
Change in Self efficacy for healthy eating and exercise | Baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  These secondary outcomes measures aim to explore the mechanisms of the intervention by assessing the "mediated effect" on the outcomes of insulin sensitivity and weight-specific QoL through the following putative mediators targeted in the program: self-efficacy for healthy eating and exercise.
Change in Social support from family and friends on healthy eating and exercise. | Baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  These secondary outcomes measures aim to explore the mechanisms of the intervention by assessing the "mediated effect" on the outcomes of insulin sensitivity and weight-specific QoL through the following putative mediators targeted in the program: Social support from family and friends on healthy eating and exercise.

OTHER OUTCOMES:
Initial incremental cost effectiveness of intervention vs. standard care | Analysis for the outcome is expected to occur approximately 4 years after the initial baseline testing. Data for analysis will be consist of one year ELSC cost.
  Analysis will be conducted on the initial incremental cost effectiveness of the intervention compared to no intervention on changes in insulin sensitivity and prevention of diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Q Shaibi, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

REFERENCES:
- [Background] Williams AN, Konopken YP, Keller CS, Castro FG, Arcoleo KJ, Barraza E, Patrick DL, Olson ML, Shaibi GQ. Culturally-grounded diabetes prevention program for obese Latino youth: Rationale, design, and methods. Contemp Clin Trials. 2017 Mar;54:68-76. doi: 10.1016/j.cct.2017.01.004. Epub 2017 Jan 16. PMID 28104469
- [Result] Soltero EG, Olson ML, Williams AN, Konopken YP, Castro FG, Arcoleo KJ, Keller CS, Patrick DL, Ayers SL, Barraza E, Shaibi GQ. Effects of a Community-Based Diabetes Prevention Program for Latino Youth with Obesity: A Randomized Controlled Trial. Obesity (Silver Spring). 2018 Dec;26(12):1856-1865. doi: 10.1002/oby.22300. Epub 2018 Nov 14. PMID 30426694
- [Result] Olson ML, Renteria-Mexia A, Connelly MA, Vega-Lopez S, Soltero EG, Konopken YP, Williams AN, Castro FG, Keller CS, Yang HP, Todd MW, Shaibi GQ. Decreased GlycA after lifestyle intervention among obese, prediabetic adolescent Latinos. J Clin Lipidol. 2019 Jan-Feb;13(1):186-193. doi: 10.1016/j.jacl.2018.09.011. Epub 2018 Sep 22. PMID 30342918
- [Result] Renteria-Mexia A, Vega-Lopez S, Olson ML, Swan PD, Lee CD, Williams AN, Shaibi GQ. Effects of a lifestyle intervention on markers of cardiometabolic risk and oxidized lipoproteins among obese adolescents with prediabetes. Public Health Nutr. 2019 Mar;22(4):706-713. doi: 10.1017/S1368980018003476. Epub 2018 Dec 27. PMID 30588900
- See also: PI's Research Webpage — http://www.public.asu.edu/~gshaibi/